CLINICAL TRIAL: NCT02289690
Title: A Phase 1 Dose Escalation and Phase 2 Randomized Double-Blind Study of Veliparib in Combination With Carboplatin and Etoposide as a Therapy of Treatment-Naïve Extensive Stage Disease Small Cell Lung Cancer
Brief Title: Dose Escalation and Double-blind Study of Veliparib in Combination With Carboplatin and Etoposide in Treatment-naive Extensive Stage Disease Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: M14-361; 2014-001764-35 (EudraCT Number)
Expanded Access: NCT03123211 (No longer available)
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Small Cell Lung Cancer
Keywords: Extensive Stage Smal Cell Lung Cancer; ABT-888; Veliparib; PARP - Poly (ADP) ribose polymerase
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — veliparib; Carboplatin; Etoposide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Phase 1 was open-label, phase 2 was conducted in a double-blind manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase 1: Veliparib + Carboplatin + Etoposide (Experimental): Participants in Phase 1 will be sequentially assigned to ascending dose levels of veliparib in combination with carboplatin/etoposide for up to four 21-day cycles.
  Participants without evidence of disease progression will continue on veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
  Interventions: Drug: Veliparib; Drug: Carboplatin; Drug: Etoposide
- Phase 2: Veliparib + Carboplatin + Etoposide -> Veliparib (Experimental): Participants will receive veliparib 240 mg in combination with carboplatin/etoposide for four to six 21-day cycles followed by veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
  Interventions: Drug: Veliparib; Drug: Carboplatin; Drug: Etoposide
- Phase 2: Veliparib + Carboplatin + Etoposide -> Placebo (Experimental): Participants will receive veliparib 240 mg in combination with carboplatin/etoposide for four to six 21-day cycles followed by placebo monotherapy continuous dosing (21-day cycles) until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: Veliparib; Drug: Carboplatin; Drug: Etoposide; Drug: Placebo
- Phase 2: Placebo + Carboplatin + Etoposide -> Placebo (Active Comparator): Participants will receive placebo in combination with carboplatin/etoposide for four to six 21-day cycles followed by placebo monotherapy continuous dosing (21-day cycles) until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Placebo

INTERVENTIONS:
Drug: Veliparib — Capsules administered orally twice a day according to the dosing schedule.
  Other Names: ABT-888
  Arms: Phase 1: Veliparib + Carboplatin + Etoposide; Phase 2: Veliparib + Carboplatin + Etoposide -> Placebo; Phase 2: Veliparib + Carboplatin + Etoposide -> Veliparib
Drug: Carboplatin — Administered by intravenous infusion on Day 1 of each 21-day cycle over approximately 30 minutes at a target area under the curve (AUC) 5 mg/mL*minute.
Drug: Etoposide — Administered by intravenous infusion on Days 1 to 3 of every 21-day cycle over approximately 60 minutes at 100 mg/m².
  Other Names: VP-16
Drug: Placebo — Placebo to veliparib administered orally twice a day according to the dosing schedule.
  Arms: Phase 2: Placebo + Carboplatin + Etoposide -> Placebo; Phase 2: Veliparib + Carboplatin + Etoposide -> Placebo

SUMMARY:
The study seeks to assess the efficacy of veliparib (ABT-888) in combination with carboplatin and etoposide in participants with extensive disease small cell lung cancer (ED SCLC).

DETAILED DESCRIPTION:
This is a Phase 1, open-label, dose-escalation/Phase 2 randomized double-blind study of veliparib in combination with carboplatin and etoposide and maintenance veliparib monotherapy.

Participants in Phase 1 will be sequentially assigned to ascending dose levels of veliparib in combination with standard carboplatin/etoposide regimen for up to four 21-day cycles based on the observed toxicities. The study design for Phase 1 will follow a traditional "3 + 3" dose-escalation protocol.

Once the veliparib recommended Phase 2 dose (RPTD) and schedule is determined, enrollment into Phase 2 will begin. Participants from the Phase 1 dose-escalation portion of the study are not eligible for enrollment into the Phase 2 portion. Participants in Phase 2 will be randomized in a 1:1:1 ratio to carboplatin, etoposide, placebo followed by placebo maintenance (Arm C), or carboplatin, etoposide, veliparib followed by either veliparib (Arm A) or placebo (Arm B) maintenance. Randomization for Phase 2 will be stratified by baseline lactate dehydrogenase (LDH) level (> upper limit of normal [ULN] vs. ≤ ULN), and gender.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with histologically or cytologically confirmed extensive-stage disease SCLC which is newly diagnosed and chemotherapy naive
2. Phase 1 ONLY: histologically or cytologically confirmed advanced/metastatic solid tumors for which carboplatin/etoposide treatment is considered appropriate.
3. Subject in Phase 2 only: must have measurable disease per RECIST 1.1.
4. Subjects with ED SCLC must consent to provide available archived formalin fixed paraffin embedded (FFPE) tissue sample of SCLC lesion (primary or metastatic) for central review and biomarker analysis.
5. Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 1.
6. Subject must have adequate hematologic, renal and hepatic function.

Exclusion Criteria:

1. Phase 1 ONLY: Subject has had any prior anti-cancer therapy other than:

   Hormonal, non-myelosuppressive, biologic, targeted, or immune therapy (must be completed ≥ 4 weeks prior to Cycle 1 Day -2).

   One line of cytotoxic chemotherapy (must be completed ≥ 4 weeks prior to Cycle 1 Day -2).

   Adjuvant/neoadjuvant radiotherapy (must be completed ≥ 12 months prior to Cycle 1 Day -2, with field not involving > 10% of bone marrow reserve).
2. Phase 2 ONLY: Subject has had any prior chemotherapy, radiotherapy, investigational anti-cancer agents or biologic therapy for the disease under study. Single non-target lesion irradiation with intent of symptom palliation is allowed if ≥ 4 weeks prior Cycle 1 Day -2.
3. Subject has current central nervous system (CNS) or leptomeningeal metastases or history of CNS or leptomeningeal metastases.
4. Subject has a history of seizures within 12 months of Cycle 1 Day-2 or diagnosed neurological condition placing subject at the increased risk of seizures.
5. Subject has received anti-cancer Chinese medicine or anti-cancer herbal remedies within 14 days prior to Cycle 1 Day-2.
6. Subject has had major surgery within 6 weeks prior to Cycle 1 Day-2 (subjects must have completely recovered from any previous surgery prior Cycle 1 Day-2).
7. Subject has clinically significant and uncontrolled major medical condition(s) including but not limited to:

   * Uncontrolled nausea/vomiting/diarrhea;
   * Active uncontrolled infection;
   * History of hepatitis B (HBV) with surface antigen (HBsAg) positivity within 3 months prior to the date of informed consent for this study (if no test has been performed within 3 months, it must be done at screening);
   * History of hepatitis C (HCV) with HCV ribonucleic acid (RNA) positivity within 3 months prior to the date of informed consent for this study (if no test has been performed within 3 months it must be done at screening);
   * Symptomatic congestive heart failure (Yew York Heart Association [NYHA] class ≥ II);
   * Unstable angina pectoris or cardiac arrhythmia (except atrial fibrillation);
   * Psychiatric illness/social situation that would limit compliance with study requirements;
   * Any other medical condition, which in the opinion of the Investigator, places the subject at an unacceptably high risk for toxicities.
8. The subject has a history of another active cancer within the past 3 years except cervical cancer in situ, in situ carcinoma of the bladder, squamous or basal cell carcinoma of the skin or another in situ cancer that is considered cured by the investigator (e.g., in situ prostate cancer, breast DCIS).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (62):
- United States (9):
  - Mayo Clinic - Scottsdale /ID# 129127, Scottsdale, Arizona
  - Univ of Colorado Cancer Center /ID# 129220, Aurora, Colorado
  - Emory University Hospital /ID# 141682, Atlanta, Georgia
  - Georgia Regents University /ID# 148567, Augusta, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 137088, Chicago, Illinois
  - Herbert Herman Cancer Center /ID# 167020, Lansing, Michigan
  - Gabrail Cancer Center Research /ID# 129216, Canton, Ohio
  - Allegheny General Hospital /ID# 147328, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center /ID# 129213, Houston, Texas
- Australia (4):
  - Southern Medical Day Care Ctr /ID# 155498, Wollongong, New South Wales
  - The Townsville Hospital /ID# 155499, Douglas, Queensland
  - Peninsula & South Eastern Haem /ID# 155497, Frankston, Victoria
  - Border Medical /ID# 157894, Wodonga, Victoria
- Belgium (5):
  - Cliniques Universitaires Saint Luc /ID# 151024, Woluwe-Saint-Lambert, Brussels Capital
  - CHU de Liege /ID# 151025, Liège, Liege
  - UZ Antwerp /ID# 151026, Edegem
  - C.H.U.de Mons Borinage /ID# 151023, Mons
  - CHU UCL Namur /ID# 151022, Namur
- Canada (4):
  - University of Calgary /ID# 152544, Calgary, Alberta
  - Cross Cancer Institute /ID# 132883, Edmonton, Alberta
  - Juravinski Cancer Clinic /ID# 152543, Hamilton, Ontario
  - Hopital du Sacre Coeur Montreal /ID# 154436, Montreal, Quebec
- Czechia (4):
  - Nemocnice Na Plesi s.r.o. /ID# 149825, Nová Ves pod Pleší, Pribram
  - Nemocnice Novy Jicin /ID# 149838, Nový Jičín
  - Vitkovicka nemocnice a. s. /ID# 149839, Ostrava
  - Multiscan s.r.o. /ID# 150887, Pardubice
- France (3):
  - CHU Dupuytren /ID# 153622, Limoges, Franche-Comte
  - Centre Hospitalier Le Mans /ID# 158103, Le Mans, Sarthe
  - Centre Hosp Intercommunal de Creteil /ID# 157970, Créteil, Val-de-Marne
- Hungary (8):
  - Orszagos Koranyi Pulmonologiai Intezet /ID# 151351, Budapest XII, Budapest
  - Markusovszky Egyetemi Oktatókórház /ID# 158806, Szombathely, Vas County
  - Debreceni Egyetem Klinikai Központ /ID# 151354, Debrecen
  - Veszprem Megyei Tudogyogyintez /ID# 158807, Farkasgyepű
  - Petz Aladar Megyei Oktato Korh /ID# 155352, Győr
  - Matrahaza Gyogyintezet /ID# 151355, Kékesteto
  - Fejer Megyei Szent Gyorgy Korh /ID# 151352, Székesfehérvár
  - Jasz-Nagykun-Szolnok Megyei /ID# 155090, Szolnok
- Netherlands (5):
  - Universitair Medisch Centrum Groningen /ID# 131252, Groningen
  - Ziekenhuis St. Jansdal /ID# 151974, Harderwijk
  - Atrium-Orbis Zuyderland Medisch Centrum /ID# 149830, Heerlen
  - Erasmus Medisch Centrum /ID# 131251, Rotterdam
  - Isala /ID# 151975, Zwolle
- Romania (3):
  - S.C. Centrul de Oncologie Sf. Nectarie S.R.L. /ID# 161137, Craiova, Dolj
  - Oncocenter Oncologie Clinica S /ID# 151694, Timișoara, Timiș County
  - S.C. Radiotherapy Center Cluj /ID# 165137, Cluj-Napoca
- Russia (7):
  - NN Blokhin Russian Cancer /ID# 152329, Moscow, Moscow
  - Sverdlovsk Regional Oncology Center Dispensary /ID# 152328, Yekaterinburg, Sverdlovsk Oblast
  - Belgorod Oncology Dispensary /ID# 152330, Belgorod
  - Univercity Headache Clynic,LTD /ID# 161708, Moscow
  - Murmansk RCH P.A. Bayandina /ID# 152331, Murmansk
  - Road Hospital Open Joint Stock Company Russian Railways /ID# 152731, Saint Petersburg
  - Ogarev Mordovia State Univ /ID# 152327, Saransk
- South Korea (4):
  - Dong-A University Hospital /ID# 153187, Busan, Busan Gwang Yeogsi
  - Chungbuk National Univ Hosp /ID# 153186, Cheongju-si
  - Chonnam National University Hwasun Hospital /ID# 153188, Jeonnam
  - Asan Medical Center /ID# 153185, Seoul
- Spain (6):
  - Hospital Stanta Creu i Sant Pau /ID# 151254, Barcelona
  - Hosp Univ Quiron Dexues /ID# 130302, Barcelona
  - Hospital Universitario Gregori /ID# 164982, Madrid
  - Hosp Univ 12 de Octubre /ID# 151252, Madrid
  - Hosp Univ Madrid Sanchinarro /ID# 130301, Madrid
  - Hosp Univ Puerta de Hierro Maj /ID# 151253, Majadahonda

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Result] Atrafi F, Groen HJM, Byers LA, Garralda E, Lolkema MP, Sangha RS, Viteri S, Chae YK, Camidge DR, Gabrail NY, Hu B, Tian T, Nuthalapati S, Hoening E, He L, Komarnitsky P, Calles A. A Phase I Dose-Escalation Study of Veliparib Combined with Carboplatin and Etoposide in Patients with Extensive-Stage Small Cell Lung Cancer and Other Solid Tumors. Clin Cancer Res. 2019 Jan 15;25(2):496-505. doi: 10.1158/1078-0432.CCR-18-2014. Epub 2018 Oct 16. PMID 30327308

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 52 study sites located in 12 countries (Australia, Belgium, Canada, Czech Republic, France, Hungary, Korea, the Netherlands, Romania, Russian Federation, Spain, United States).
Pre-assignment Details: Participants in Phase 1 were sequentially assigned to ascending dose levels of veliparib in combination with standard carboplatin/etoposide regimen. Participants in Phase 2 were randomized equally to placebo, carboplatin/etoposide followed by placebo maintenance, or to veliparib, carboplatin/etoposide followed by veliparib or placebo maintenance.
Groups:
- Phase 1: Veliparib 80 mg BID 7 Days + Carboplatin/Etoposide: Participants received 80 mg veliparib orally twice a day (BID) on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 5 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered intravenously (IV) on Day 1 at a target area under the curve (AUC) 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 120 mg BID 7 Days + Carboplatin/Etoposide: Participants received 120 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 5 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 160 mg BID 7 Days + Carboplatin/Etoposide: Participants received 160 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 5 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 200 mg BID 7 Days + Carboplatin/Etoposide: Participants received 200 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 5 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 240 mg BID 7 Days + Carboplatin/Etoposide: Participants received 240 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 5 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 240 mg BID 14 Days + Carboplatin/Etoposide: Participants received 240 mg veliparib orally BID on Days -2 to 12 (14 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 12 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 240 mg BID 21 Days + Carboplatin/Etoposide: Participants received 240 mg veliparib orally BID on Days -2 to Day 19 (continuous schedule) in combination with carboplatin/etoposide for up to four 21-day cycles. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib: Participants received veliparib 240 mg BID on Day -2 to 12 (14-day schedule), carboplatin AUC 5 mg/mL*min administered on Day 1, and etoposide 100 mg/m² administered on Days 1 to 3 of each 21-day cycle for up to 6 cycles.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo: Participants received veliparib 240 mg BID on Day -2 to 12 (14-day schedule), carboplatin AUC 5 mg/mL*min administered on Day 1, and etoposide 100 mg/m² administered on Days 1 to 3 of each 21-day cycle for up to 6 cycles.
  Participants without evidence of disease progression received placebo monotherapy BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Phase 2: Placebo + Carboplatin/Etoposide -> Placebo: Participants received placebo BID on Day -2 to 12 (14-day schedule), carboplatin AUC 5 mg/mL*min on Day 1, and etoposide 100 mg/m² on Days 1 to 3 of each 21-day cycle for up to 6 cycles.
  Participants without evidence of disease progression received placebo monotherapy BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase 1: Veliparib 80 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 120 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 160 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 200 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 14 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 21 Days + Carboplatin/Etoposide | Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib | Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo | Phase 2: Placebo + Carboplatin/Etoposide -> Placebo
Started | 4 | 3 | 4 | 3 | 8 | 14 | 4 | 61 | 59 | 61
Received Study Drug | 4 | 3 | 4 | 3 | 8 | 14 | 4 | 60 | 58 | 60
Completed (Completed indicates participants remaining on study.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 4 | 3 | 8 | 14 | 4 | 61 | 59 | 61
Not completed — Adverse Event Related to Progression | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 2
Not completed — Progressive Disease, Per Protocol | 3 | 2 | 3 | 2 | 5 | 13 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 49 | 45 | 41
Not completed — Sponsor Discontinued Study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 7 | 15
Not completed — Other | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Veliparib 80 mg BID 7 Days + Carboplatin/Etoposide: Participants received 80 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 5 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered intravenously (IV) on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 160 mg BID 7 Days + Carboplatin/Etoposide: Participants received 160 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 5 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease pParticipants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Veliparib 80 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 120 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 160 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 200 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 14 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 21 Days + Carboplatin/Etoposide | Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib | Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo | Phase 2: Placebo + Carboplatin/Etoposide -> Placebo | Total
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 8 | 14 | 4 | 61 | 59 | 61 | 221
Age, Continuous [Median (Full Range); unit: years] — Population: Phase 1 and Phase 2 were analyzed separately.
  years
    Phase 1: number analyzed (Participants) | 4 | 3 | 4 | 3 | 8 | 14 | 4 | 0 | 0 | 0 | 40
    Phase 1 | 74.0 [55.0 to 79.0] | 69.0 [62.0 to 75.0] | 62.5 [56.0 to 74.0] | 54.0 [52.0 to 68.0] | 52.0 [43.0 to 63.0] | 66.0 [52.0 to 72.0] | 59.0 [57.0 to 62.0] |  |  |  | 62.5 [43.0 to 79.0]
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 59 | 61 | 181
    Phase 2 |  |  |  |  |  |  |  | 62.0 [39.0 to 77.0] | 64.0 [46.0 to 86.0] | 63.0 [37.0 to 87.0] | 63.0 [37.0 to 87.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 1 | 2 | 5 | 1 | 21 | 21 | 23 | 79
  Male | 1 | 3 | 2 | 2 | 6 | 9 | 3 | 40 | 38 | 38 | 142
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 3 | 4 | 3 | 8 | 14 | 4 | 55 | 51 | 52 | 198
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 4
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7 | 7 | 18
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis.
  0 = Fully Active (Most Favorable Activity);
  1. = Restricted activity but ambulatory;
  2. = Ambulatory but unable to carry out work activities;
  3. = Limited Self-Care;
  4. = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 - Fully active | 1 | 1 | 1 | 1 | 2 | 3 | 2 | 21 | 16 | 23 | 71
    1 - Restricted but ambulatory | 3 | 2 | 3 | 2 | 5 | 11 | 1 | 39 | 42 | 37 | 145
    Missing | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as any of the following drug-related toxicities, graded according to the Common Toxicity Criteria for Adverse Events (CTCAE), V.4.0:
  1. Events associated with treatment delay >14 days in initiating Cycle 2 therapy:
     Grade 4 thrombocytopenia, neutropenia, or febrile neutropenia, or Grade 3 febrile neutropenia with fever for > 7 days
  2. Grade ≥ 3 non-hematologic toxicity with ≥ 2 grade increase from baseline and attributed to veliparib treatment, excluding nausea or vomiting for ≤ 48 hours or inadequately treated, electrolyte abnormalities resolving in ≤ 24 hours, hypersensitivity reactions or alopecia
  3. Grade 2 non-hematologic toxicity of ≥ 2 grade increase from baseline, attributed to veliparib treatment requiring delay of >14 days in initiation of Cycle 2
  4. Any toxicity of ≥ 2-grade increase from baseline, attributed to veliparib and requiring a dose modification in Cycle 1 or omission of carboplatin, >1 daily etoposide dose, or >30% veliparib doses in Cycle 1
Time Frame: Cycle 1 Day -2 to pre-dose on Cycle 2 Day 1 (23 days)
Population: Phase 1 participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Veliparib 80 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 120 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 160 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 200 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 14 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 21 Days + Carboplatin/Etoposide
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 8 | 14 | 4
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Phase 1: Veliparib 80 mg BID 7 Days + Carboplatin/Etoposide vs Phase 1: Veliparib 120 mg BID 7 Days + Carboplatin/Etoposide vs Phase 1: Veliparib 160 mg BID 7 Days + Carboplatin/Etoposide vs Phase 1: Veliparib 200 mg BID 7 Days + Carboplatin/Etoposide vs Phase 1: Veliparib 240 mg BID 7 Days + Carboplatin/Etoposide vs Phase 1: Veliparib 240 mg BID 14 Days + Carboplatin/Etoposide vs Phase 1: Veliparib 240 mg BID 21 Days + Carboplatin/Etoposide; A primary objective of Phase 1 was to establish the recommended phase 2 dose (RP2D) for veliparib combined with carboplatin and etoposide. The RP2D was determined by the rate of DLTs and overall tolerability of veliparib plus carboplatin and etoposide; Test type: Other; RP2D for veliparib in mg BID for 14 days = 240 — The RP2D for veliparib was determined to be 240 mg BID for 14 days with carboplatin (AUC 5 mg/mL*min) on Day 1 and etoposide (100 mg/m²) on Days 1 to 3 during 21-day cycles for 4 cycles

2. Primary Outcome: Phase 1: Maximum Observed Plasma Concentration (Cmax) of Veliparib
Description: Plasma concentrations of veliparib were determined using a validated online solid-phase extraction followed by high-performance liquid chromatography with tandem mass spectrometric detection (HPLC LC-MS/MS). The lower limit of quantitation (LLOQ) for veliparib was established at ≥ 1.05 ng/mL.
Time Frame: Cycle 1 Day 1 predose and at 1, 2, 3, 5, 8, and 24 hours post-dose
Population: Phase 1 participants who were administered at least 1 dose of study drug, had at least 1 reported PK sample concentration and for whom Cmax could be calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Phase 1: Veliparib 80 mg BID + Carboplatin/Etoposide: Participants received 80 mg veliparib orally twice a day (BID) on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles. Carboplatin was administered intravenously (IV) on Day 1 at a target area under the curve (AUC) 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
- Phase 1: Veliparib 120 mg BID + Carboplatin/Etoposide: Participants received 120 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
- Phase 1: Veliparib 160 mg BID + Carboplatin/Etoposide: Participants received 160 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
- Phase 1: Veliparib 200 mg BID + Carboplatin/Etoposide: Participants received 200 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
- Phase 1: Veliparib 240 mg BID + Carboplatin/Etoposide: Participants received 240 mg veliparib orally BID (Days -2 to 5 for 7-day schedule, Days -2 to 12 for 14-day schedule or Days -2 to 19 for continuous dosing) in combination with carboplatin/etoposide for up to four 21-day cycles. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
Arm/Group | Phase 1: Veliparib 80 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 120 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 160 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 200 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID + Carboplatin/Etoposide
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 22
μg/mL | 0.620 (17) | 1.00 (31) | 1.39 (29) | 1.44 (10) | 1.99 (25)

3. Primary Outcome: Phase 1: Time to Maximum Observed Plasma Concentration (Tmax) of Veliparib
Description: as for outcome 2
Time Frame: Cycle 1 Day 1 predose and at 1, 2, 3, 5, 8, and 24 hours post-dose
Population: Phase 1 participants who were administered at least 1 dose of study drug, had at least 1 reported PK sample concentration and for whom Tmax could be calculated.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: Veliparib 80 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 120 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 160 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 200 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID + Carboplatin/Etoposide
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 22
hours | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]

4. Primary Outcome: Phase 1: Area Under the Plasma Concentration-time Curve From Time 0 to 8 Hours Post-dose (AUC[0-8]) of Veliparib
Description: The area under the plasma concentration-time curve from time 0 to 8 hours post-dose for veliparib was estimated using non-compartmental methods.
Time Frame: Cycle 1 Day 1 predose and at 1, 2, 3, 5, 8, and 24 hours post-dose
Population: Phase 1 participants who were administered at least 1 dose of study drug, had at least 1 reported PK sample concentration and for whom AUC(0-8) could be calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Phase 1: Veliparib 80 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 120 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 160 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 200 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID + Carboplatin/Etoposide
Number analyzed (Participants) | 4 | 3 | 4 | 2 | 22
μg*h/mL | 3.18 (14) | 4.24 (25) | 7.51 (28) | 6.66 (4) | 9.29 (37)

5. Primary Outcome: Phase 1: Area Under the Plasma Concentration-time Curve From Time 0 to 12 Hours Post-dose (AUC[0-12]) of Veliparib
Description: The area under the plasma concentration-time curve from time 0 to 12 hours post-dose for veliparib was estimated using non-compartmental methods. AUC(0-12) was calculated by assuming the concentration at 12 hours post-dose was the same as the pre-dose concentration.
Time Frame: Cycle 1 Day 1 predose and at 1, 2, 3, 5, 8, and 24 hours post-dose
Population: Phase 1 participants who were administered at least 1 dose of study drug, had at least 1 reported PK sample concentration and for whom AUC(0-12) could be calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Phase 1: Veliparib 80 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 120 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 160 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 200 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID + Carboplatin/Etoposide
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 22
μg*h/mL | 4.07 (15) | 5.25 (27) | 9.71 (31) | 8.35 (6) | 11.6 (40)

6. Primary Outcome: Phase 1: Dose-normalized Maximum Observed Plasma Concentration of Veliparib
Description: Plasma concentrations of veliparib were determined using a validated online solid-phase extraction followed by high-performance liquid chromatography with tandem mass spectrometric detection (HPLC LC-MS/MS). The lower limit of quantitation (LLOQ) for veliparib was established at ≥ 1.05 ng/mL.
  Dose normalized Cmax is calculated as Cmax / veliparib dose in mg.
Time Frame: Cycle 1 Day 1 predose and at 1, 2, 3, 5, 8, and 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/mg
Arm/Group | Phase 1: Veliparib 80 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 120 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 160 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 200 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID + Carboplatin/Etoposide
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 22
(ng/mL)/mg | 7.75 (16) | 8.35 (31) | 8.66 (29) | 7.19 (10) | 8.31 (25)

7. Primary Outcome: Phase 1: Dose-normalized Area Under the Plasma Concentration-time Curve From Time 0 to 8 Hours Post-dose of Veliparib
Description: The area under the plasma concentration-time curve from time 0 to 8 hours post-dose for veliparib was estimated using non-compartmental methods. Dose normalized AUC(0-8) is calculated as AUC(0-8) / veliparib dose in mg.
Time Frame: Cycle 1 Day 1 predose and at 1, 2, 3, 5, 8, and 24 hours post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h/mL)/mg
Arm/Group | Phase 1: Veliparib 80 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 120 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 160 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 200 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID + Carboplatin/Etoposide
Number analyzed (Participants) | 4 | 3 | 4 | 2 | 22
(ng*h/mL)/mg | 39.8 (14) | 35.3 (25) | 46.9 (28) | 33.3 (4) | 38.7 (37)

8. Primary Outcome: Phase 1: Dose-normalized Area Under the Plasma Concentration-time Curve From Time 0 to 12 Hours Post-dose of Veliparib
Description: The area under the plasma concentration-time curve from time 0 to 12 hours post-dose for veliparib was estimated using non-compartmental methods. AUC(0-12) was calculated by assuming the concentration at 12 hours post-dose was the same as the pre-dose concentration. Dose normalized AUC(0-12) is calculated as AUC(0-12) / veliparib dose in mg.
Time Frame: Cycle 1 Day 1 predose and at 1, 2, 3, 5, 8, and 24 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h/mL)/mg
Arm/Group | Phase 1: Veliparib 80 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 120 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 160 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 200 mg BID + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID + Carboplatin/Etoposide
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 22
(ng*h/mL)/mg | 50.9 (15) | 43.8 (27) | 60.7 (31) | 41.7 (6) | 48.5 (40)

9. Primary Outcome: Phase 1: Maximum Observed Plasma Concentration (Cmax) of Etoposide With and Without Veliparib
Description: Etoposide plasma concentrations were determined using liquid chromatography with tandem mass spectrometric detection with a lower limit of quantitation 160 ng/mL.
Time Frame: Cycle 1 Day 1 (coadministered with veliparib and carboplatin), and on Cycle 2 Day 1 (co-administered with carboplatin but in the absence of veliparib) at 55 minutes (5 minutes before the end of infusion) and 3, 5, 8, and 24 hours post-dose.
Population: Phase 1 participants who received at least 1 dose of study drug, had at least 1 reported PK concentration for each time point and for whom Cmax could be calculated. Participants in the Veliparib 240 mg BID 21-day (continuous) dosing group and participants whose etoposide dose was reduced in Cycle 2 are not included in the Cycle 2 Day 1 analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Etoposide Cycle 1 Day 1 (With Veliparib): Phase 1 participants received 100 mg/m² etoposide intravenously with carboplatin target AUC 5.0 mg*min/mL and veliparib 80 to 240 mg BID on Cycle 1 Day 1.
- Etoposide Cycle 2 Day 1 (No Veliparib): Phase 1 participants received etoposide 100 mg/m² and carboplatin target AUC 5.0 mg*min/mL on Day 1 of Cycle 2. No veliparib was administered.
Arm/Group | Etoposide Cycle 1 Day 1 (With Veliparib) | Etoposide Cycle 2 Day 1 (No Veliparib)
Number analyzed (Participants) | 37 | 23
μg/mL | 16.9 (18) | 16.4 (21)

10. Primary Outcome: Phase 1: Time to Maximum Observed Plasma Concentration (Tmax) of Etoposide With and Without Veliparib
Description: as for outcome 9
Time Frame: as for outcome 9
Population: Phase 1 participants who received at least 1 dose of study drug, had at least 1 reported PK concentration for each time point and for whom Tmax could be calculated. Participants in the Veliparib 240 mg BID 21-day (continuous) dosing group are not included in the Cycle 2 Day 1 analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Etoposide Cycle 1 Day 1 (With Veliparib) | Etoposide Cycle 2 Day 1 (No Veliparib)
Number analyzed (Participants) | 37 | 28
hours | 0.9 [0.8 to 3.0] | 0.9 [0.9 to 3.7]

11. Primary Outcome: Phase 1: Area Under the Concentration-time Curve From Time 0 to Time of Last Measurable Concentration (AUC[0-t]) of Etoposide With and Without Veliparib
Description: The area under the plasma concentration-time curve from 0 to the last measurable concentration (24 hours) of etoposide was estimated using using non-compartmental methods.
Time Frame: as for outcome 9
Population: Phase 1 participants who received at least 1 dose of study drug, had at least 1 reported PK concentration for each time point and for whom AUC could be calculated. Participants in the Veliparib 240 mg BID 21-day (continuous) dosing group and participants whose etoposide dose was reduced in Cycle 2 are not included in the Cycle 2 Day 1 analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Etoposide Cycle 1 Day 1 (With Veliparib) | Etoposide Cycle 2 Day 1 (No Veliparib)
Number analyzed (Participants) | 35 | 22
μg*h/mL | 102 (23) | 94.7 (18)

12. Primary Outcome: Phase 1: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC[0-∞]) of Etoposide With and Without Veliparib
Description: The area under the plasma concentration-time curve from 0 to infinity for etoposide was estimated using using non-compartmental methods.
Time Frame: as for outcome 9
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | Etoposide Cycle 1 Day 1 (With Veliparib) | Etoposide Cycle 2 Day 1 (No Veliparib)
Number analyzed (Participants) | 35 | 22
μg*h/mL | 112 (56) | 99.5 (18)

13. Primary Outcome: Phase 1: Terminal Phase Elimination Half-life (t1/2) of Etoposide With and Without Veliparib
Description: The terminal half-life of etoposide was estimated using using non-compartmental methods. Values reported represent the harmonic mean ± pseudo-standard deviation.
Time Frame: as for outcome 9
Population: Participants in Phase 1 who received at least 1 dose of study drug and had at least 1 reported PK sample concentration for each time point and for whom t1/2 could be calculated. Participants in the Veliparib 240 mg BID 21-day (continuous) dosing group are not included in the Cycle 2 Day 1 analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Etoposide Cycle 1 Day 1 (With Veliparib) | Etoposide Cycle 2 Day 1 (No Veliparib)
Number analyzed (Participants) | 35 | 27
hours | 5.7 (1.5) | 5.0 (1.2)

14. Primary Outcome: Phase 1: Dose-normalized Maximum Observed Plasma Concentration (Cmax) of Etoposide With and Without Veliparib
Description: Etoposide plasma concentrations were determined using liquid chromatography with tandem mass spectrometric detection with a lower limit of quantitation 160 ng/mL. Dose normalized Cmax is calculated as Cmax / etoposide dose in mg/m².
Time Frame: as for outcome 9
Population: Phase 1 participants who received at least 1 dose of study drug, had at least 1 reported PK concentration for each time point and for whom Cmax could be calculated. Participants in the Veliparib 240 mg BID 21-day (continuous) dosing group are not included in the Cycle 2 Day 1 analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/(mg/m²)
Arm/Group | Etoposide Cycle 1 Day 1 (With Veliparib) | Etoposide Cycle 2 Day 1 (No Veliparib)
Number analyzed (Participants) | 37 | 28
(ng/mL)/(mg/m²) | 169 (18) | 170 (20)

15. Primary Outcome: Phase 1: Dose-normalized Area Under the Concentration-time Curve From Time 0 to Time of Last Measurable Concentration (AUC[0-t]) of Etoposide With and Without Veliparib
Description: The area under the plasma concentration-time curve from 0 to the last measurable concentration (24 hours) of etoposide was estimated using using non-compartmental methods. Dose normalized AUC(0-t) is calculated as AUC(0-t) / etoposide dose in mg/m².
Time Frame: as for outcome 9
Population: Phase 1 participants who received at least 1 dose of study drug, had at least 1 reported PK concentration for each time point and for whom AUC could be calculated. Participants in the Veliparib 240 mg BID 21-day (continuous) dosing group are not included in the Cycle 2 Day 1 analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h/mL)/(mg/m²)
Arm/Group | Etoposide Cycle 1 Day 1 (With Veliparib) | Etoposide Cycle 2 Day 1 (No Veliparib)
Number analyzed (Participants) | 35 | 27
(ng*h/mL)/(mg/m²) | 1020 (23) | 952 (21)

16. Primary Outcome: Phase 1: Dose-normalized Area Under the Concentration-time Curve From Time 0 to Infinity (AUC[0-∞]) of Etoposide With and Without Veliparib
Description: The area under the plasma concentration-time curve from 0 to infinity for etoposide was estimated using using non-compartmental methods. Dose normalized AUC(0-∞) is calculated as AUC(0-∞) / etoposide dose in mg/m².
Time Frame: as for outcome 9
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h/mL)/(mg/m²)
Arm/Group | Etoposide Cycle 1 Day 1 (With Veliparib) | Etoposide Cycle 2 Day 1 (No Veliparib)
Number analyzed (Participants) | 35 | 27
(ng*h/mL)/(mg/m²) | 1120 (56) | 1020 (20)

17. Primary Outcome: Phase 2: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time from the date of randomization to the date of earliest radiographic disease progression or death provided no radiographic disease progression occurred.
  If a participant did not have an event of disease progression and had not died on or prior to the cutoff for PFS analysis, the participant's data was censored at the date of their last disease assessment or randomization date provided participant did not have any post-baseline disease assessment.
  Disease assessments were performed using computed tomography according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
  Progressive Disease (PD) was defined as at least a 20% increase in the size of target lesions and an absolute increase of at least 5 mm taking as reference the smallest lesion size recorded since the treatment started (baseline or after), or the appearance of one or more new lesions.
Time Frame: From randomization up to the date the 126th PFS event was reached; Median time on follow-up was 7.3, 7.1, and 8.9 months in each treatment group respectively.
Population: All participants randomized in Phase 2
Measure: Median (80% Confidence Interval); unit: months
Groups:
- Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib: Participants in Arm A received veliparib 240 mg BID on Day -2 to 12 (14-day schedule), carboplatin AUC 5 mg/mL*min administered on Day 1, and etoposide 100 mg/m² administered on Days 1 to 3 of each 21-day cycle for up to 6 cycles.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo: Participants in Arm B received veliparib 240 mg BID on Day -2 to 12 (14-day schedule), carboplatin AUC 5 mg/mL*min administered on Day 1, and etoposide 100 mg/m² administered on Days 1 to 3 of each 21-day cycle for up to 6 cycles.
  Participants without evidence of disease progression received placebo monotherapy BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
- Phase 2: Placebo + Carboplatin/Etoposide -> Placebo: Participants in Arm C received placebo BID on Day -2 to 12 (14-day schedule), carboplatin AUC 5 mg/mL*min on Day 1, and etoposide 100 mg/m² on Days 1 to 3 of each 21-day cycle for up to 6 cycles.
  Participants without evidence of disease progression received placebo monotherapy BID continuous dosing (21-day cycles) until disease progression or unacceptable toxicity.
Arm/Group | Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib | Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo | Phase 2: Placebo + Carboplatin/Etoposide -> Placebo
Number analyzed (Participants) | 61 | 59 | 61
months | 5.8 [5.6 to 6.8] | 5.7 [5.6 to 5.8] | 5.6 [5.1 to 6.7]
Statistical Analysis 1: Comparison: Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib vs Phase 2: Placebo + Carboplatin/Etoposide -> Placebo; The primary efficacy analysis in the Phase 2 portion of the study was the comparison of PFS among participants who received veliparib in combination with carboplatin and etoposide followed by veliparib maintenance monotherapy (Arm A) vs. placebo in combination with carboplatin and etoposide followed by placebo maintenance monotherapy (Arm C). Statistical significance was determined by a two-sided p-value ≤ 0.2; Test type: Superiority; p = 0.059, Log Rank; Two-sided log-rank test stratified by lactate dehydrogenase (LDH) level; Hazard Ratio (HR) = 0.665, 80% CI 2-sided [0.503 to 0.880] — Hazard ratio estimate was obtained from a Cox proportional hazards model stratified by LDH level. A hazard ratio < 1 favors veliparib in combination with carboplatin and etoposide followed by veliparib maintenance monotherapy (Arm A)
Statistical Analysis 2: Comparison: Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo vs Phase 2: Placebo + Carboplatin/Etoposide -> Placebo; If the primary analysis of PFS (Arm A vs Arm C) was statistically significant a fixed sequence testing procedure was to be performed with a 2-sided significance level of 0.2 for the following key secondary endpoints: 1. OS (Arm A vs Arm C) 2. PFS (Arms B vs Arm C) 3. OS (Arm B vs Arm C) 4. ORR (Arm A vs Arm C) 5. ORR (Arm B vs Arm C) If significance versus Arm C was not demonstrated, all endpoints later in the testing hierarchy were to be considered exploratory; Test type: Superiority; p = 0.924, Log Rank; Two-sided log-rank test stratified by lactate dehydrogenase (LDH) level; Hazard Ratio (HR) = 0.979, 80% CI 2-sided [0.744 to 1.288] — Hazard ratio estimate was obtained from a Cox proportional hazards model stratified by LDH level. A hazard ratio of < 1 favors veliparib in combination with carboplatin and etoposide followed by placebo maintenance monotherapy (Arm B)

18. Secondary Outcome: Phase 2: Overall Survival
Description: Overall survival (OS) is defined as the time from the date of randomization to the date of death. If a participant did not die on or prior to the cut-off for OS analysis, the participant's data were censored at the date of their last known alive date, which is defined as the last date of the last survival follow-up visit, the start date of the last AE, the start date or end date of the last dose of any study drugs, the last lab and vital sign collection date, or the last disease assessment date, whichever occurred last.
Time Frame: From randomization until the end of study; median time on follow-up was 10.0, 8.6, and 11.7 months in each treatment group respectively.
Population: All participants randomized in Phase 2
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib | Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo | Phase 2: Placebo + Carboplatin/Etoposide -> Placebo
Number analyzed (Participants) | 61 | 59 | 61
months | 10.1 [9.2 to 11.4] | 10.0 [8.0 to 12.7] | 12.4 [11.1 to 13.6]
Statistical Analysis 1: Comparison: Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib vs Phase 2: Placebo + Carboplatin/Etoposide -> Placebo; [analysis description as in outcome 17, analysis 2]; Test type: Superiority; p = 0.088, Log Rank; Two-sided log rank test stratified by LDH level; Hazard Ratio (HR) = 1.432, 80% CI 2-sided [1.092 to 1.879] — Hazard ratio estimate was obtained from a Cox proportional hazards model stratified by LDH level. A hazard ratio of < 1 favors veliparib in combination with carboplatin and etoposide followed by veliparib maintenance monotherapy (Arm A)
Statistical Analysis 2: Comparison: Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo vs Phase 2: Placebo + Carboplatin/Etoposide -> Placebo; [analysis description as in outcome 17, analysis 2]; Test type: Superiority; p = 0.083, Log Rank; Two-sided log rank test stratified by LDH level; Hazard Ratio (HR) = 1.460, 80% CI 2-sided [1.104 to 1.931] — [estimate comment as in outcome 17, analysis 2]

19. Secondary Outcome: Phase 2: Objective Response Rate
Description: Objective response rate (ORR) is defined as the percentage of participants with objective response (confirmed) as assessed by the investigator using RECIST version 1.1. Objective response includes both complete response (CR) and partial response (PR). Response must be confirmed at a subsequent tumor assessment at least 28 days apart. Participants with no post-baseline confirmed response were counted as non-responders.
  CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. No new lesions.
  PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, and no new lesions.
Time Frame: Tumor assessments were performed every 6 weeks for the first 30 weeks and every 9 weeks thereafter until disease progression; median time on follow-up was 7.3, 7.1, and 8.9 months in each group respectively.
Population: All participants randomized in Phase 2
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib | Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo | Phase 2: Placebo + Carboplatin/Etoposide -> Placebo
Number analyzed (Participants) | 61 | 59 | 61
percentage of participants | 77.0 [68.7 to 84.0] | 59.3 [50.1 to 68.0] | 63.9 [55.0 to 72.2]
Statistical Analysis 1: Comparison: Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib vs Phase 2: Placebo + Carboplatin/Etoposide -> Placebo; [analysis description as in outcome 17, analysis 2]; Test type: Superiority; p = 0.115, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by LDH level; Odds Ratio (OR) = 1.9, 80% CI 2-sided [1.1 to 3.2] — Odds ratio was from a Cochran-Mantel-Haenszel test stratified by LDH level. An odds ratio of > 1 favors veliparib in combination with carboplatin and etoposide followed by veliparib maintenance monotherapy (Arm A)
Statistical Analysis 2: Comparison: Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo vs Phase 2: Placebo + Carboplatin/Etoposide -> Placebo; [analysis description as in outcome 17, analysis 2]; Test type: Superiority; p = 0.604, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by LDH level; Odds Ratio (OR) = 0.8, 80% CI 2-sided [0.5 to 1.3] — Odds ratio was from a Cochran-Mantel-Haenszel test stratified by LDH level. An odds ratio of > 1 favors veliparib in combination with carboplatin and etoposide followed by placebo maintenance monotherapy (Arm B)

20. Secondary Outcome: Phase 1: Number of Participants With Adverse Events
Description: The intensity of each adverse event (AE) was assessed utilizing the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0, and according to the following: Grade 1 (Mild): AE is transient and easily tolerated by the participant; Grade 2 (Moderate): AE causes the participant discomfort and interrupts the participant's usual activities; Grade 3/4 (Severe): The adverse event causes considerable interference with the participant's usual activities and may be incapacitating or life-threatening; Grade 5: Death.
  Serious adverse events were those that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization, resulted in congenital anomaly, or persistent or significant disability/incapacity.
Time Frame: From first dose of any study drug to 30 days after the last dose; the median duration of treatment with veliparib across all groups in Phase 1 was 127.5 days.
Population: Participants in Phase 1 who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Veliparib 80 mg BID 7 Days + Carboplatin/Etoposide: Participants received 80 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 5 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered intravenously (IV) on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg twice a day until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 120 mg BID 7 Days + Carboplatin/Etoposide: Participants received 120 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 5 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 160 mg BID 7 Days + Carboplatin/Etoposide: Participants received 160 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 5 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 200 mg BID 7 Days + Carboplatin/Etoposide: Participants received 200 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 5 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 240 mg BID 7 Days + Carboplatin/Etoposide: Participants received 240 mg veliparib orally BID on Days -2 to 5 (7 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 5 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 240 mg BID 14 Days + Carboplatin/Etoposide: Participants received 240 mg veliparib orally BID on Days -2 to 12 (14 days) in combination with carboplatin/etoposide for up to four 21-day cycles, with the exception of Cycle 2, when veliparib was administered on Days 2 to 12 to allow for evaluation of potential impact of veliparib on etoposide pharmacokinetics. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID until disease progression or unacceptable toxicity.
- Phase 1: Veliparib 240 mg BID 21 Days + Carboplatin/Etoposide: Participants received 240 mg veliparib orally BID on Days -2 to Day 19 (continuous schedule) in combination with carboplatin/etoposide for up to four 21-day cycles. Carboplatin was administered IV on Day 1 at a target AUC 5 mg/mL*minute and etoposide 100 mg/m² IV on Days 1 to 3 of every 21-day cycle.
  Participants without evidence of disease progression continued on veliparib monotherapy at 400 mg BID until disease progression or unacceptable toxicity.
Arm/Group | Phase 1: Veliparib 80 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 120 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 160 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 200 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 14 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 21 Days + Carboplatin/Etoposide
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 8 | 14 | 4
Participants
  Any adverse event | 4 | 3 | 4 | 3 | 8 | 14 | 4
  Any AE Grade 3/4 | 4 | 3 | 4 | 3 | 7 | 14 | 4
  Any serious adverse event | 3 | 1 | 3 | 2 | 3 | 6 | 3
  Any fatal adverse event | 0 | 0 | 1 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to the end of study, maximum time on follow-up was 26 months. Treatment-emergent adverse events and serious adverse events were collected from first dose of study drug until 30 days after the last dose of study drug; Maximum duration of treatment in Phase 1 was 541 days and maximum duration of treatment in Phase 2 was 654 days.
Description: All-cause mortality is reported for all participants enrolled in Phase 1 and randomized in Phase 2. Adverse events are reported for all participants who received at least 1 dose of study drug.
Arm/Group | Phase 1: Veliparib 80 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 120 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 160 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 200 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 7 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 14 Days + Carboplatin/Etoposide | Phase 1: Veliparib 240 mg BID 21 Days + Carboplatin/Etoposide | Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib | Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo | Phase 2: Placebo + Carboplatin/Etoposide -> Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 1/4 | 1/3 | 0/8 | 0/14 | 0/4 | 50/61 | 45/59 | 41/61
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/3 | 3/4 | 2/3 | 3/8 | 6/14 | 3/4 | 33/60 | 39/58 | 27/60
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 4/4 | 3/3 | 8/8 | 14/14 | 4/4 | 57/60 | 53/58 | 53/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Veliparib 80 mg BID 7 Days + Carboplatin/Etoposide (N=4) | Phase 1: Veliparib 120 mg BID 7 Days + Carboplatin/Etoposide (N=3) | Phase 1: Veliparib 160 mg BID 7 Days + Carboplatin/Etoposide (N=4) | Phase 1: Veliparib 200 mg BID 7 Days + Carboplatin/Etoposide (N=3) | Phase 1: Veliparib 240 mg BID 7 Days + Carboplatin/Etoposide (N=8) | Phase 1: Veliparib 240 mg BID 14 Days + Carboplatin/Etoposide (N=14) | Phase 1: Veliparib 240 mg BID 21 Days + Carboplatin/Etoposide (N=4) | Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib (N=60) | Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo (N=58) | Phase 2: Placebo + Carboplatin/Etoposide -> Placebo (N=60)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 2 (3)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 7 (7) | 3 (3)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 2 (2)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (9) | 2 (2)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIABETES INSIPIDUS (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
PALATAL OEDEMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DISEASE PROGRESSION (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SUDDEN CARDIAC DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUDDEN DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IMPLANT SITE CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
ORCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLEURAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 3 (3) | 1 (1)
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA LEGIONELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
VASCULAR PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 5 (6) | 5 (5)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MOTOR DYSFUNCTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TOXIC NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
AORTITIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL EMBOLISM (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VENA CAVA THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Veliparib 80 mg BID 7 Days + Carboplatin/Etoposide (N=4) | Phase 1: Veliparib 120 mg BID 7 Days + Carboplatin/Etoposide (N=3) | Phase 1: Veliparib 160 mg BID 7 Days + Carboplatin/Etoposide (N=4) | Phase 1: Veliparib 200 mg BID 7 Days + Carboplatin/Etoposide (N=3) | Phase 1: Veliparib 240 mg BID 7 Days + Carboplatin/Etoposide (N=8) | Phase 1: Veliparib 240 mg BID 14 Days + Carboplatin/Etoposide (N=14) | Phase 1: Veliparib 240 mg BID 21 Days + Carboplatin/Etoposide (N=4) | Phase 2: Veliparib + Carboplatin/Etoposide -> Veliparib (N=60) | Phase 2: Veliparib + Carboplatin/Etoposide -> Placebo (N=58) | Phase 2: Placebo + Carboplatin/Etoposide -> Placebo (N=60)
ANAEMIA (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 2 (9) | 1 (3) | 4 (11) | 7 (18) | 2 (6) | 35 (104) | 35 (105) | 26 (55)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 7 (15) | 12 (27) | 3 (13)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 2 (8) | 0 (0) | 4 (11) | 8 (34) | 2 (6) | 36 (94) | 33 (86) | 28 (71)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 3 (6) | 5 (16) | 1 (3) | 22 (58) | 23 (62) | 12 (22)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (1)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTOTOXICITY (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLINDNESS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EYE IRRITATION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE PAIN (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LACRIMATION INCREASED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITREOUS DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 3 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (3) | 2 (2) | 0 (0) | 2 (2)
ANAL INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 14 (17) | 13 (19) | 11 (15)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 7 (11) | 1 (1) | 8 (11) | 11 (21) | 11 (12)
DIVERTICULUM (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 7 (8) | 2 (3) | 4 (5)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERUCTATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 3 (3)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (4) | 2 (7) | 2 (4) | 5 (8) | 9 (16) | 1 (1) | 29 (57) | 23 (47) | 21 (29)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
ORAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCTITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETCHING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 3 (4) | 2 (2) | 3 (4)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (4) | 1 (2) | 1 (2) | 2 (3) | 1 (1) | 13 (20) | 10 (12) | 8 (9)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (8) | 0 (0) | 9 (16) | 11 (26) | 2 (3)
CHEST PAIN (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
CREPITATIONS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CRYING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FACE OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 2 (3) | 3 (5) | 1 (2) | 2 (4) | 6 (6) | 9 (20) | 1 (1) | 15 (23) | 16 (17) | 10 (12)
FEELING ABNORMAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEELING COLD (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
INJECTION SITE EXTRAVASATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE HAEMATOMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE PHLEBITIS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOSS OF CONTROL OF LEGS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
NECROSIS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
OEDEMA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (3) | 6 (7) | 5 (5)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 3 (3)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 6 (9) | 2 (2) | 8 (10)
SWELLING (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SWELLING FACE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HEPATIC PAIN (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 4 (4) | 0 (0)
ORAL FUNGAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 3 (3)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
CHEMICAL PHLEBITIS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL HEADACHE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 3 (6) | 2 (10)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 5 (6) | 3 (4) | 2 (3)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (3)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HLA MARKER STUDY POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (5) | 1 (1) | 1 (2) | 1 (2) | 6 (20) | 2 (8) | 1 (2) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (11) | 1 (3) | 1 (2) | 1 (6) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINE OUTPUT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 5 (13) | 0 (0) | 3 (3) | 2 (2) | 7 (11)
WEIGHT INCREASED (Investigations) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 1 (5) | 1 (2) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (3) | 2 (4) | 3 (3) | 0 (0) | 3 (5) | 7 (16) | 2 (2) | 17 (20) | 12 (14) | 14 (16)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 6 (7)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (6)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (3) | 5 (5) | 9 (13) | 7 (8)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 4 (5) | 1 (1) | 10 (24) | 7 (9) | 9 (12)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 6 (8) | 7 (7) | 4 (5)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (4) | 0 (0) | 6 (8) | 2 (6) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 6 (6) | 0 (0) | 9 (11) | 7 (7) | 9 (9)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
COCCYDYNIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 3 (7) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (8) | 4 (4)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 1 (2) | 4 (4) | 2 (2)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TENDON PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ATAXIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
DIZZINESS (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 3 (6) | 2 (2) | 5 (6) | 9 (13) | 3 (4)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 4 (6) | 2 (2)
HEAD DISCOMFORT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 10 (11) | 9 (11) | 7 (7)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
MUSCLE CONTRACTIONS INVOLUNTARY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEVICE OCCLUSION (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 7 (11) | 1 (1) | 4 (5) | 5 (6) | 4 (4)
RESTLESSNESS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST MICTURITION DRIBBLE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY HESITATION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
PERINEAL PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 5 (6) | 2 (2) | 6 (6) | 5 (5) | 7 (7)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 5 (5) | 2 (2) | 12 (16) | 9 (11) | 7 (10)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 2 (2)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 3 (3)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (4)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (3) | 2 (2) | 3 (5) | 8 (12) | 1 (3) | 22 (27) | 17 (19) | 18 (20)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PIGMENTATION DISORDER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 2 (2)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STICKY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 2 (2) | 1 (3) | 3 (3)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-11-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT02289690/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT02289690/SAP_001.pdf